CLINICAL TRIAL: NCT02071693
Title: Cholinergic Pathways Hyperintensities Scale Could Not Predict the Change of Cognitive Status of Parkinson's Disease Patients After Bilateral STN DBS.
Brief Title: A Retrospective Study of the Relationship Between White Matter Hyperintensities(WMHs) Within the Cholinergic Pathways and the Cognition of PD Patients After Bilateral STN DBS
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chen Ling, Doctor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: [2008] 20; 2010B080701107 (Other Grant/Funding Number: Guangdong Science and Technology Foundation)
Record Dates: First submitted 2014-02-23; First posted 2014-02-26 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Parkinson's Disease
Keywords: subthalamic nucleus; deep brain stimulation; cognition; white matter hyperintensities
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To retrospectively investigate the relationship between the Cholinergic Pathways Hyperintensities Scale (CHIPS) score and the change of cognitive status of Parkinson's disease (PD) patients after bilateral subthalamic nucleus deep brain stimulation (STN DBS).

DETAILED DESCRIPTION:
In this observational study, we will retrospectively analyze 38 PD patients who received bilateral STN DBS in the First Affiliated Hospital of Sun Yat-sen University during the year of 2008-2012. All patients will be evaluated by Unified Parkinson's Disease Rating Scale part III(UPDRSIII) before and after operation. Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment(MoCA) in the on medication condition pre-operation and on stimulation on medication condition post-operation. The follow-up time points are one week pre-operation and 6, 12, 24 months post-operation. Before operation, white matter hyperintensities（WMHs）in the cholinergic pathways will be determined on a 3.0 Tesla MRI, using the visual rating scale of Cholinergic Pathways Hyperintensities Scale (CHIPS). A correlation analysis will be conducted to investigate the relationship between CHIPS score and the change of cognitive status of PD patients after bilateral STN DBS retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease according to United Kingdom Parkinson's Disease Brain Bank Criteria
* Experience bilateral STN DBS surgery in the First Affiliated Hospital, Sun Yat-sen University, China.
* Preoperative 3.0 Tesla MRI scanning.

Exclusion Criteria:

* Loss to follow-up
* Participation in other clinical trials

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients treated with bilateral STN DBS in the First Affiliated Hospital during the year of 2008-2012.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change of MoCA score during follow-up and its relationship with preoperative CHIPS score | Pre-operation and 6, 12, 24 months post-operation
Change of MMSE score during follow-up and its relationship with preoperative CHIPS score | Pre-operation and 6, 12, 24 months post-operation

SECONDARY OUTCOMES:
Change of UPDRS III score during follow-up and its relationship with preoperative CHIPS score | Pre-operation and 6, 12, 24 months post-operation

CONTACTS AND LOCATIONS:
Overall Officials: Ling Chen, MD,PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China